CLINICAL TRIAL: NCT04707365
Title: Interactions Between Tumor, Tumor Microenvironment and Immune System in Digestive Cancers : Impact on Survival and Response to Treatment
Brief Title: Microenvironment and Immunity of Digestive Cancers - East Paris Multicentric Cohort
Acronym: MICADO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP190090; IDRCB :2019-A00071-56 (Other: ANSM)
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer; Pancreas Tumor; Biliary Tract Tumor; Immune System and Related Disorders
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Retrospective and prospective monocentric cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- digestive cancers (Experimental): Colorectal and pancreatobiliary cancers
  Interventions: Biological: Tumor samples

INTERVENTIONS:
Biological: Tumor samples — for each patient: liver sampling, blood samples ( serum, plasma, PBMC, whole blood), per-endoscopic bile sampling, stool samples, and materials derived from fresh tumors

SUMMARY:
Colorectal and pancreatobiliary cancers are the most common digestive cancers. Their incidence has particularly increased over the last few decades, leading to suspicion that environmental factors are involved. In addition, strategies for the therapeutic management of these cancers are evolving in the context of the development of immunotherapies.

Tumor microenvironment is a potential source of new diagnostic, prognostic and predictive markers and new therapeutic targets. The links between tumor microenvironment and modulation of the immune system in colorectal and pancreatobiliary cancers are poorly understood. Molecular classifications have been proposed for these cancers, but their link with immunity and response to treatment remains to be explored.

Objective : explore links between molecular subtypes, tumor microenvironment, host (immune system, pre-metastatic niche, intestinal microbiota, metabolism), and survival (prognostic value), response (predictive value) and tolerance (toxicities) to treatments in digestive cancers, in particular colorectal and pancreatobiliary cancers.

Method: Retrospective and prospective monocentric cohort study

ELIGIBILITY:
Inclusion Criteria:

* Colorectal or pancreatic adenocarcinoma or biliary tract adenocarcinoma
* Cytologically or histologically proven adenocarcinoma, regardless of stage and treatment
* Age ≥ 18 years old
* Diagnosed from 2015 onwards
* Signed Consent
* Affiliation to a social security scheme (including CMU (Universal health coverage))

Exclusion Criteria:

* Patient under guardianship, curatorship or safeguarding of justice
* Pregnant or breastfeeding woman
* Any medical, psychological or social situation that could prevent compliance with the protocol according to the investigator's assessment.
* Refusal to participate in the study
* Patient on AME (state medical assistance)
* Persons deprived of liberty by a judicial or administrative decision
* Persons under psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2035-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
overall survival | observation from first cancer treatment date until date of death or 10 years follow up if patient alive
  Overall survival (OS): vital status (alive/deceased)

CONTACTS AND LOCATIONS:
Overall Officials: Pr Tournigand, Study Director — AP-HP Henri Mondor Créteil

IPD SHARING:
Plan to Share IPD: No
AP-HP is the owner of the data and no use or transmission to a third party may be made without its prior consent.